CLINICAL TRIAL: NCT04655781
Title: Displacement of the Retina After Idiopathic Macular Hole Surgery With Different Internal Limiting Membrane Peeling Patterns
Brief Title: Internal Limiting Membrane Peeling on Retinal Displacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILM Peeling
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Internal Limiting Membrane Peeling
Keywords: Retinal displacement; Idiopathic macular hole; Internal limiting membrane peeling
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-T group (Experimental): ILM was peeled off from nasal retina to temporal retina.
  Interventions: Procedure: idiopathic macular hole (MH) surgery
- T-N group (Experimental): ILM was peeled off from temporal retina to nasal retina
  Interventions: Procedure: idiopathic macular hole (MH) surgery

INTERVENTIONS:
Procedure: idiopathic macular hole (MH) surgery — Idiopathic Macular Hole Surgery with Different Internal Limiting Membrane Peeling Patterns

SUMMARY:
The purpose of this study is to investigate displacement of the retina after idiopathic macular hole surgery with different internal limiting membrane peeling patterns.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. All patients with idiopathic MH will be randomly allocated into two groups, N-T group or T-N group.

ELIGIBILITY:
Inclusion Criteria:

Eyes with idiopathic macular hole

Exclusion Criteria:

Eyes having re-do macular hole surgery, with high myopia, with proliferative vitreoretinopathy or with a retinal detachment combined with the MH, with other macular diseases, such as age-related macular degeneration.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
T-OD | preoperation to postoperative 6 months
  measurement of temporal vessel to optic disc

IPD SHARING:
Plan to Share IPD: No